CLINICAL TRIAL: NCT00656383
Title: Effectiveness and Efficiency of Two Models of Delivering Care to a Chronic Wound Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: The Ottawa Hospital (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Margaret Harrison, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOP-42497
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Varicose Ulcer
Keywords: venous ulcer, leg ulcer, stasis ulcer
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Client is randomized to receive leg ulcer treatment in the home
  Interventions: Other: Clients receive leg ulcer care in their homes
- 2 (Active Comparator): Client randomized to receive leg ulcer care in the clinic
  Interventions: Other: Clients randomized to nurse-led clinic

INTERVENTIONS:
Other: Clients randomized to nurse-led clinic — Clients receive leg ulcer care in a nurse-led clinic; both groups are treated by the same health care providers using the same protocol
  Other Names: Usual Care; Best Practice; Venous Leg Ulcer treatment
  Arms: 2
Other: Clients receive leg ulcer care in their homes — Clients receive leg ulcer care in at home; both groups are treated by the same health care providers using the same protocol
  Other Names: Leg Ulcer Care; Usual Care; Best Practice
  Arms: 1

SUMMARY:
Individuals referred to home care for leg ulcer management were randomized to nurse home visits (usual care) or nurse-run community clinics (intervention). The primary outcome will be the time to healing rates at three months. Secondary outcomes are: time to healing of all ulcers within the 12 month follow-up period, time to first recurrence of a healed ulcer, the number of weeks patients were free from ulcers, function, pain, and health related quality of life, client and provider satisfaction. We hypothesize that nurse-run neighborhood clinics result in better healing rates, more cost-effective care, and improved client and provider satisfaction than the home visiting model.

DETAILED DESCRIPTION:
The management of chronic wounds in the community is a pressing issue for home care authorities. The care of leg ulcers represents a considerable expense to the health care system. It has been estimated that the care of venous leg ulcers alone consumes 1% of the national health care budgets of the UK and France. A one-month prevalence study in the Ottawa Carleton region (pop. 750,000) revealed that 126 Community Care Access Centre Clients (CCAC - the regional health care authority) received over 1500 home nursing visits. During the course of a year this represents more than $600,000 in home nursing visits for this condition in just one Ontario region. There is evidence supporting effective wound management but this is not necessarily what patients receive. As well, appropriate evidence-based, efficient, community-based care must be supported by ready access to specialized facilities. Research from other countries suggest that reorganization of services which includes nurse-run clinic care near to home, evidence-based protocols, and enhanced linkages with secondary and tertiary services may result in improvements in healing rates and reductions in expenditures. These international studies provide optimism that with reorganization of care within the Canadian context we can deliver community services for improved outcomes. However, only with a rigorous evaluation of the effectiveness and efficiency can we understand if such changes in the Canadian context are beneficial.

Objective:

To evaluate the effectiveness and efficiency of two models of service delivery: traditional single service delivery model (home visiting) compared to nurse-led community clinics.

Research Questions:

1. What are the health outcomes (healing, function, plain and quality of life) for two models of care (nurse-run neighbourhood clinics vs. home care) for the population with leg ulcers?
2. What are health services utilization and expenditures associated with the two models of care?
3. What is client and provider satisfaction with the nurse-run neighbourhood clinics and home nursing care?
4. What are the barriers and supports to implementing neighbourhood leg ulcer clinics?

Study Design and Method:

A randomized health services controlled trial of nurse-run neighbourhood leg ulcer clinics (intervention) and home care (current practice) with a cost-effectiveness analysis. A repeated measures design will be used to assess healing and ulcer improvement, quality of life and patient satisfaction over time.

Outcome measures:

The primary outcome measure is the proportion of limbs healed by three months. Secondary outcome measures are: time to complete healing, ulcer size, ulcer recurrence, function, pain, quality of life, client and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

The client:

* Admission to home care for care of a venous leg ulcer (below the knee to the foot)
* Ability to travel to clinic
* No major contraindication for clinic care (eg not being able to leave an ill spouse, refusal, etc.)

Exclusion Criteria:

* Treatment is contraindicated
* The ulcer in question is not venous
* The client cannot travel outside the home or travel is impeded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2000-10; Primary Completion 2004-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Proportion in each study arm of ulcerated limbs completely healed at 3 months | 3 months

SECONDARY OUTCOMES:
Time to complete healing, ulcer size, and ulcer recurrence over 12 months | 12 months
Client function, pain and health-related quality of life | 12 months
Client and provider satisfaction | 12 months
Health services expenditure and utilization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaret B Harrison, RN, PhD, Principal Investigator — The Ottawa Hospital; Ian D Graham, PhD, Study Director — Clinical Epidemiology Unit, Ottawa Hospital-Civic Campus; Philip S Wells, PhD, Study Director — The Ottawa Hospital; Susan VanDeVelde, PhD, Study Director — Victorian Order of Nurses, Ottawa-Carleton Branch; Judith L Threinen, BSR, MHA, Study Director — Ottawa-Carleton Community Care Access Centre; Donna I Nicholson, Dip O&A, Study Director — Ottawa Carleton Community Care Access Centre
Locations (2):
- Canada (2):
  - Ottawa Carleton Community Care Access Centre, Ottawa, Ontario
  - Victorian Order of Nurses, Ottawa-Carleton, Ottawa, Ontario

REFERENCES:
- [Derived] Harrison MB, Graham ID, Lorimer K, Vandenkerkhof E, Buchanan M, Wells PS, Brandys T, Pierscianowski T. Nurse clinic versus home delivery of evidence-based community leg ulcer care: a randomized health services trial. BMC Health Serv Res. 2008 Nov 26;8:243. doi: 10.1186/1472-6963-8-243. PMID 19036149